CLINICAL TRIAL: NCT01782079
Title: Assessment of Probiotic Lactobacillus Brevis CD2 Strain Persistence in Oral Cavity. A Pilot Study
Brief Title: L. Brevis CD2 Strain Persistence in Oral Cavity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Luciana Mosca, PhD, Principal Investigator, University of Roma La Sapienza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LB - 001
Record Dates: First submitted 2013-01-18; First posted 2013-02-01 (Estimated); Last update posted 2013-03-25 (Estimated); Status verified 2013-03

CONDITIONS: Oral Health
Keywords: Lactobacillus brevis; Oral health; Bacterial adhesion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- L. brevis (Experimental)
  Interventions: Dietary Supplement: L. brevis

INTERVENTIONS:
Dietary Supplement: L. brevis

SUMMARY:
The aim of this study is to select the optimal conditions for quantification in the oral cavity of Lactobacillus brevis CD2, a probiotic strain contained in a commercially available dietary supplement and to assess its persistency after oral administration. Different sets of primers for L. brevis detection will be tested in real-time PCR reactions to find optimal amplification efficiency and target specificity. Primers ability in the identification of L. brevis DNA will be assessed in a pilot study conducted on 12 healthy volunteers clinically free of oral pathologies. The subjects will take 3 tablets/day for 3 days and one tablet on the 4th day. Clinical samples (dorsal surface of tongue, first molar, vestibular fornix and saliva) will be collected at baseline (before beginning the trial), at T0 (in the morning before the assumption of the last tablet) and 3, 6, and 9 hours after taking the last tablet. The quantities of L. brevis DNA will be compared to the total number of bacteria present in the samples. The activity of the enzyme arginine deiminase, responsible for oral pH homeostasis (particularly abundant in the CD2 strain) will be also assessed in the saliva samples before and after treatment, by HPLC measurements.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Healthy subjects with no oral cavity pathologies
* Written informed consent

Exclusion Criteria:

* Patients with oral diseases
* Patients with systemic diseases
* Celiac patients or subjects affected by allergic reactions to soy proteins
* Use of antibiotics or other probiotics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Quantification and persistency of Lactobacillus brevis CD2 after oral administration | 4 days
  Mucosal surface colonization in various mouth sites will be assessed by measuring the number of bacteria by Real Time PCR. Quantities of L. brevis DNA will be compared to the total number of bacteria present in the samples.

SECONDARY OUTCOMES:
Arginine deiminase activity | 4 days
  Enzyme activity, measured as the amount of citrulline formed per minute in the assay conditions, will be determined in saliva samples by HPLC measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Università La Sapienza, Roma, Italy